CLINICAL TRIAL: NCT04408859
Title: Quality of Life in Patient With Neoadjuvant Chemotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Gastric Cancer
Brief Title: Quality of Life in Advanced Gastric Cancer Patients Receiving Neoadjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Xiangqian Su, Chief of GI surgery IV, Peking University Cancer Hospital & Institute
Other Study IDs: QOL-201804
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: QOL; Quality of Life;Gastric Cancer; Gastrectomy;Neoadjuvant Chemotherapy
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NACS: The patients with advanced gastric cancer who received neoadjuvant chemotherapy followed by surgery（NACS）.
  Interventions: Drug: Neoadjuvant Chemotherapy
- SA: The patients with advanced gastric cancer who received surgery alone.

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy — The patients receive neoadjuvant chemotherapy for 2-4 cycles before surgery.
  Groups: NACS

SUMMARY:
The purpose of this study is to explore the influence of neoadjuvant chemotherapy in the long term quality of life with advanced gastric cancer patients.

DETAILED DESCRIPTION:
Preoperative adjuvant chemotherapy combined with postoperative adjuvant therapy mode was included in the 2018 version of the National Comprehensive Cancer Network (NCCN) guideline as an optional treatment (category 2B) for prospective resectable advanced gastric cancer cases (≥cT2, any N).At home and abroad, the research on neoadjuvant chemotherapy for advanced gastric cancer mainly focuses on the safety and long-term survival, and there are few studies on the quality of life. This study, according to EORTC QLQ-C30 and QLQ-STO22 assessment scale, explores the long term effect of neoadjuvant chemotherapy on the quality of life in patients with advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients age older than 18 years (including 18 years old);
* Diagnosis of adenocarcinoma of the stomach
* The clinic stage is ≥T2 and any N stage
* Patient had curative surgical resection, including proximal, distal, or total gastrectomy

Exclusion Criteria:

* Psychiatric or psychological abnormality precluding informed consent or ability to complete questionnaires
* Non-psychiatric disorder causing a lack of capacity to give consent or an inability to complete questionnaires (ie dementia, stroke)
* Early gastric cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had curative resection at Beijing Cancer Hospital for advanced gastric cancer and finish the questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2022-01-10 (Estimated); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life index | 2 years
  The change of quality of life index during the 2 years after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No